CLINICAL TRIAL: NCT00965055
Title: Atorvastatin vs. Atorvastatin/Ezetimibe in Patients With Hypo-response to Initial Dose Statin Therapy
Brief Title: Ezetimibe in Patients Hypo-responsive to Statins
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated due to inability to recruit subjects. A total of 2/100 anticipated were radomized.
Sponsor: University of California, San Diego (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Ori Ben-Yehuda, Professor of Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 090948
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Results first posted 2019-08-21 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: High Cholesterol; Coronary Artery Disease
MeSH Terms: conditions — Hypercholesterolemia; Coronary Artery Disease | interventions — Ezetimibe; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atorvastatin (Placebo Comparator)
  Interventions: Drug: Atorvastatin
- Atorvastatin/Ezetimibe (Experimental)
  Interventions: Drug: Ezetimibe; Drug: Atorvastatin

INTERVENTIONS:
Drug: Ezetimibe — 10 mg
  Other Names: Zetia; Lipitor
  Arms: Atorvastatin/Ezetimibe
Drug: Atorvastatin — Visit 1: (atorvastatin open label challenge): Those who complete the initial screening and washout period will receive open label atorvastatin 10 mg daily for 6 weeks to verify compliance and confirm hyporesponse to statin therapy.
  Visit 2: After 6 weeks of therapy repeat baseline fasting cholesterol. Those with LDL-c reduction of 25% or less will be able to proceed to next phase. Patients with greater than 25% LDL-C reduction will be excluded. We expect to randomize 80 patients
  Visit 2a: Dispensing of first randomized drug allocation- all patients receive open label atorvastatin 10 mg with additional ezetimibe 10 mg or matching placebo. No blood test during this visit.
  Visit 3, 4, 5: Dose titration to atorvastatin to 20 mg, 40 mg, 80 mg, respectively, after fasting blood test
  Blood collected in visits 3, 4, and 5 will be stored for additional tests regarding cholesterol metabolism and inflammation.
  Visit 6: Final cholesterol panel and conclusion of study period

SUMMARY:
Response to statin therapy for elevated low density lipoprotein is variable and may be influenced by cholesterol absorption. This study will evaluate whether combination therapy with atorvastatin/ezetimibe will be superior to atorvastatin alone in subjects who have less than 25% LDL reduction on starting dose statin (eg, atorvastatin 10 mg daily or simvastatin 20 mg daily).

DETAILED DESCRIPTION:
Specific Aim 1 To identify a patient population seen in the University of California, San Diego general internal medicine and cardiology subspecialty clinics as well as referrals from community physicians who are hyporesponsive to statin therapy (defined as an initial LDL reduction of <25% in response to 10mg of atorvastatin or 20mg of simvastatin- expected mean reduction is 35% -37% for starting dose simvastatin and atorvastatin).

Specific Aim 2 To test the hypothesis, with a prospective study, that a hyporesponse to statin therapy may be related to increased cholesterol absorption, and that this hyporesponse may be overcome by the addition of ezetimibe, a specific cholesterol absorption inhibitor.

Specific Aim 3 To evaluate whether patients with less than 25% LDL reduction on 10 mg of atorvastatin (or 20 mg of simvastatin) would achieve significantly greater LDL reduction with combination therapy (atorvastatin/ezetimibe) than with statin dose titration (using atorvastatin).

ELIGIBILITY:
Inclusion Criteria:

* Patients will need to have an LDL-C level of 130 mg/dl or greater without treatment.
* They must have demonstrated an initial LDL-C reduction of less than 25% on 10 mg of atorvastatin or 20 mg of simvastatin.
* Eligible patients will be those deemed by their physicians to be eligible for lipid lowering therapy with a statin and to have stable CAD, CAD equivalent per NCEP guidelines, or Framingham risk of 10-20%.

Exclusion Criteria:

* Recent (<3 months) diagnosis of Acute Coronary Syndromes due to ethical considerations [10].
* Pregnant patients, those planning to become pregnant, or those who are breast feeding, those with liver disease, history allergic reaction to any agent used in the trial, history of myositis, myopathy, pancreatitis, hypertriglyceridemia (TG > 400 mg/dL), history of significant alcohol or drug abuse, history of organ transplantation, or patient refusal.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-09; Primary Completion 2011-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ori Ben-Yehuda, MD, Principal Investigator — UCSD
Locations (1):
- UCSD Medical Center in Hillcrest Clinical Trials Facility, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Study Participants
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Study was not analyzed as only 2 subjects were enrolled and the study was terminated due to lack of enrollment.
Arm/Group | All Study Participants
Number analyzed (Participants) | 0
Age, Categorical
Sex: Female, Male

OUTCOME MEASURES:

1. Primary Outcome: LDL-C Reduction
Description: Study was not analyzed as only 2 subjects were enrolled and the study was terminated due to lack of enrollment.
Time Frame: 6 weeks
Population: Study was not analyzed as only 2 subjects were enrolled and the study was terminated due to lack of enrollment.
Arm/Group | All Study Participants
Number analyzed (Participants) | 0

2. Secondary Outcome: LDL-C Reduction as Well as Changes in TG, HDL, and Non-HDL Cholesterol.
Time Frame: 24 weeks
Population: Study was not analyzed as only 2 subjects were enrolled and the study was terminated due to lack of enrollment.
Arm/Group | All Study Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | All Study Participants
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
Study was not analyzed as only 2 subjects were enrolled and the study was terminated due to lack of enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes